CLINICAL TRIAL: NCT00952991
Title: A Double Blind, Cross Over, Placebo Controlled, Multiple-dose Study to Evaluate the Effects of LAF237 on Gastric Emptying, Gastric Volume and Satiety in Patients With Type 2 Diabetes.
Brief Title: The Effects of LAF237 on Gastric Function in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1721-04
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: LAF237 = vildagliptin

SUMMARY:
Administration of the incretin hormone, Glucagon-Like-Peptide-1 (GLP-1), has been shown to enhance insulin secretion and suppress glucagon secretion in response to meal ingestion. In addition, GLP-1 also delays gastric emptying and has been shown to enhance gastric accommodation. These characteristics make GLP-1 an ideal therapy for type 2 diabetes (T2D). However, because of its rapid breakdown by dipeptidylpeptidase IV (DPP IV), GLP-1 has to be administered by continuous intravenous infusion. This would be a drawback in clinical usage. LAF237 is a synthetic inhibitor of DPP IV which has been shown to raise GLP-1 levels and potentiate meal-induced insulin secretion and glucagon suppression. However, the effects of LAF237 on gastric emptying and satiety are at present unknown. The investigators propose to study the effects of LAF237 on gastric emptying, gastric volume and satiety in patients with T2D in addition to examining the direct and indirect (mediated via insulin and glucagon) of this compound on postprandial glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes without microvascular or macrovascular complications treated with diet or up to 2 oral agents

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Gastric Emptying
Gastric accommodation
Satiety
Gastrointestinal Symptoms

SECONDARY OUTCOMES:
Meal Appearance Rate
Glucose Disappearance
Endogenous Glucose Production
Insulin Secretion
Glucagon Secretion

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States